CLINICAL TRIAL: NCT02730741
Title: Study of the Efficacy and Tolerance of Oral Treatment of Lcr Restituo® Sachets (Lactobacillus Rhamnosus Lcr35®) on Intolerance to Metformin (Diarrhoea) in Patients With Diabetes Type 2
Brief Title: Study of the Efficacy and Tolerance of Oral Treatment With a Total Freeze-dried Culture of Lcr Restituo® Sachets (Lactobacillus Rhamnosus Lcr35®) on Intolerance to Metformin (Diarrhoea) in Patients With Diabetes Type 2
Acronym: PROVAME
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biose (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO_2014-02; 2014-003670-16 (EudraCT Number)
Record Dates: First submitted 2016-03-30; First posted 2016-04-06 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Antidiarrhoea
Keywords: diarrhoea; metfomin; type 2 diabetes; microbiota
MeSH Terms: conditions — Diarrhea; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lcr restituo® sachet and placebo (Experimental): The active treatment (Total freeze-dried culture of Lcr restituo® sachet) at a rate of 2 sachets of 1.5 grams per day (one sachet in the morning and one in the evening) and the placebo at a rate of 2 sachets of 1.5 grams per day (one sachet in the morning and one in the evening).
  Interventions: Drug: Lcr restituo® sachet; Drug: Placebo
- Lcr restituo® sachet (Experimental): The active treatment (Total freeze-dried culture of Lcr restituo® sachet) at a rate of 4 sachets of 1.5 grams per day (two sachets in the morning and two in the evening).
  Interventions: Drug: Lcr restituo® sachet
- Placebo (Placebo Comparator): The placebo at a rate of 4 sachets of 1.5 grams per day (two sachets in the morning and two in the evening).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lcr restituo® sachet — symptomatic treatment of diarrhoea
  Other Names: Bacilor
  Arms: Lcr restituo® sachet; Lcr restituo® sachet and placebo
Drug: Placebo
  Arms: Lcr restituo® sachet and placebo; Placebo

SUMMARY:
The mechanisms of diarrhoea under metformin are poorly known. Recent data indicate that a change in gut flora might be responsible for this intestinal disorder. The effect of metformin on the gut flora has been extensively described. It has been shown that the therapeutic effect of metformin depends on the microbiota. In agreement with these data, a recent publication has shown that metformin's main site of action in humans was the intestine. In light of these results, it now seems plausible that metformin's effect on the gut flora is responsible not only for its therapeutic effect but also for its undesirable digestive effects. In this respect, Lactobacillus rhamnosus has shown anti-diarrhoeal effects (approximately 50% reduction in diarrhoeas) in the contexts of infection-caused dysbiosis and post-antibiotic dysbiosis.

Hypothesis: Taking into account the favourable effect on intestinal dysbiosis-induced diarrhoeas observed with Lactobacillus rhamnosus, we put forward the hypothesis that Lactobacillus rhamnosus Lcr35® will have a favourable effect on metformin-induced diarrhoea.

DETAILED DESCRIPTION:
There is a diabetes pandemic: The number of diabetes patients is expected to reach 500 million worldwide by 2030, of which 90% suffering from type 2 diabetes.

Therapeutically, metformin remains the only recommended first-line treatment. However, the common digestive effects of this molecule, concerning 30 to 50% of patients, are a major obstacle to its prescription. The availability of a treatment preventing these unwanted effects would optimise the treatment of millions of diabetes patients. This would represent a considerable advantage in terms of public health due to the expected reduction in cardiovascular morbidity.

The mechanisms of diarrhoea under metformin are poorly known. Recent data indicate that a change in gut flora might be responsible for this intestinal disorder. Recent data indicate that a change in gut flora might be responsible for this intestinal disorder. The effect of metformin on the gut flora has been extensively described. It has been shown that the therapeutic effect of metformin depends on the microbiota. In agreement with these data, a recent publication has shown that metformin's main site of action in humans was the intestine. In light of these results, it now seems plausible that metformin's effect on the gut flora is responsible not only for its therapeutic effect but also for its undesirable digestive effects. In this respect, Lactobacillus rhamnosus has shown anti-diarrhoeal effects (approximately 50% reduction in diarrhoeas) in the contexts of infection-caused dysbiosis and post-antibiotic dysbiosis.

Hypothesis: Taking into account the favourable effect on intestinal dysbiosis-induced diarrhoeas observed with Lactobacillus rhamnosus, we put forward the hypothesis that Lactobacillus rhamnosus Lcr35® will have a favourable effect on metformin-induced diarrhoea.

ELIGIBILITY:
Inclusion Criteria:

Disease-related

* Patients who, from a metabolic perspective, could benefit from metformin treatment, namely patients for whom the latest available hemoglobin glycated (HbA1c) is no older than 3 months, and higher that suggested in recommendations, and lower than 9%.
* Patients with type 2 diabetes who have not received metformin treatment for at least 2 months, or treated with a non-optimal dose of metformin, i.e. 1500 mg/day or less, due to a history of diarrhoea-type digestive intolerance reported with this drug.
* Patients who at the time of entering the study have a blood sugar self-monitoring device.
* Patients whose kidney function, evaluated in reference to creatinine clearance calculated using the Cockcroft formula, is 45ml/min or higher.

Cohort-related:

* Patients aged between 18 and 75 years
* For women of childbearing age:

  * to have a negative urine pregnancy test,
  * and use a contraceptive method deemed effective by the investigator throughout the trial
* Patient able to speak and read French, having been informed of the study, and having voluntarily signed an Informed Consent Form
* Patient covered by a social security scheme

Exclusion Criteria:

Disease-related:

* Patient presenting with cardinal signs of diabetes
* Patients presenting with chronic diarrhoea or with a history of chronic intestinal inflammatory disease or having presented with an episode of acute diarrhoea in the 10 days preceding the inclusion.

Treatment-related:

* Patients presenting with a contraindication to metformin treatment other than diarrhoea-type digestive intolerance manifestations.
* Patients treated with a Inhibitors of dipeptidyl peptidase 4 (DPP-IV inhibitor).
* Patients who presented with a serious adverse event associated with metformin prescription.
* Patients who have taken orlistat in the preceding month or who have taken antibiotics in the preceding month.
* Patients who have taken probiotics in the month preceding the inclusion visit.
* Patients who have taken prebiotics in the 15 days preceding the inclusion visit.
* Patients who have an allergy to one of the active ingredients or one of the excipients in the study product.

Cohort-related:

* Patient with no referring physician.
* Patient deemed by the investigator as unable to participate in the study
* Patient unable to comply with the constraints of the protocol.
* Patient whose metabolic condition does not justify the initiation or dose increase of metformin treatment.
* History of bariatric surgery.
* Patient is immunodeficient, or has a chronic viral infection with the hepatitis B or C, or the human immunodeficiency virus (HIV virus)
* Patient is pregnant, planning a pregnancy, or without contraception.
* Breastfeeding patient.
* Patient with a previous illness which, according to the investigator, is likely to interfere with the study results or expose the patient to an additional risk.
* Patient linguistically unable (unable to speak or write French) or mentally unable to understand and sign the Informed Consent Form.
* Patient deprived of their liberty by order of the Courts or civil authorities or subject to a guardianship order.
* Patient who is likely to not comply with treatment.
* Patient unable to be contacted in the case of an emergency.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Compare number of treated patients who have had diarrhoea in the verum group and in the placebo group between Visit 2 and Visit 5. Diarrhoea evaluated using the Bristol stool scale (types 5 to 7) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Pr. Jacques MOREAU, Principal Investigator — Digestive unit - Hôpital RANGUEIL - Toulouse teaching hospital (CHU) France
Locations (1):
- BIOSE, Aurillac, France